CLINICAL TRIAL: NCT06391203
Title: A Randomised Controlled Trial to Evaluate Long-term Drainage for Patients Undergoing Decompressive Craniectomy With the Complication of Subdural Diffusion
Brief Title: Study on the Efficacy of Long-term Drainage of Subdural Effusion After Decompressive Craniectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Zhujiang Hospital (Other); Clinical Research Institute, Shanghai Jiao Tong University School of Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRAINAGE
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Brain Injury; Decompressive Craniectomy; Subdural Effusion
MeSH Terms: conditions — Brain Injuries, Traumatic; Subdural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long-term Drainage (Experimental): The drainage catheter is indwelling continuously and keeps to drainage for 7 days.
  Interventions: Procedure: Long-term Drainage
- Short-term Drainage (Active Comparator): The drainage catheter is indwelling continuously and keeps to drainage for 2 days.
  Interventions: Procedure: Short-term Drainage

INTERVENTIONS:
Procedure: Long-term Drainage — After drilling or puncture, the drainage catheter is indwelling continuously and keeps to drainage for 7 days. Keep incision sterility, record the daily fluid drainage flow, and perform biochemical and bacterial culture identification tests for CSF regularly. Removing drainage catheter when the allocated time is reached. If there is still unabsorbed effusion after the allocated time is reached, the catheter placement time is extended and the relevant information is recorded.
  Arms: Long-term Drainage
Procedure: Short-term Drainage — After drilling or puncture, the drainage catheter is indwelling continuously and keeps to drainage for 2 days. Keep incision sterility, record the daily fluid drainage flow, and perform biochemical and bacterial culture identification tests for CSF regularly. Removing drainage catheter when the allocated time is reached. If there is still unabsorbed effusion after the allocated time is reached, the catheter placement time is extended and the relevant information is recorded.
  Arms: Short-term Drainage

SUMMARY:
Drilling or puncture drainage is commonly used in TBI patients with subdural effusion following decompressive craniectomy who fail to respond to conservative treatment, but there is no exact regulation or guideline recommendation for the drainage time. The investigators aimed to conduct a randomized controlled trial to evaluate the efficacy and safety of long-term versus short-term drainage in the treatment of subdural effusion after decompressive craniectomy in patients with traumatic brain injury.

DETAILED DESCRIPTION:
Subdural effusion is a common complication following decompressive craniectomy for TBI (traumatic brain injury), with an overall incidence of 20%-50%. The clinical symptoms of subdural effusion are mainly related to the volume of effusion, and patients with a small volume of effusion may have no obvious symptoms. The flap bulge and tension of the decompression window can be seen on the same side of the decompressive craniectomy window. The specific clinical manifestations can include headache, dizziness, vomiting, epilepsy, hemiplegia, disturbance of consciousness, and other related symptoms. The degree of disturbance of consciousness changes, which can seriously affect the prognosis of patients. Drilling or puncture drainage is often used in patients with subdural effusion who fail to treat conservatively, but the drainage time has not been defined or recommended by guidelines. At present, short-term drainage is the main treatment, but there are problems such as difficulty completely absorbing the effusion or repeated recurrence. Long-term drainage can improve the absorption rate of effusion, but there is a risk of intracranial infection and other complications. Therefore, it is rarely used in clinical practice, and its clinical risks and benefits are not yet clear. Therefore, the investigators aimed to conduct a randomized controlled trial to evaluate the efficacy and safety of long-term drainage and short-term drainage in the treatment of subdural effusion after decompressive craniectomy in patients with traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral DC surgery was performed on TBI patients after injury;
2. Subdural effusion occurred for the first time and occurred within 30 days after DC surgery;
3. Unilateral effusion accumulation (can appear on the same or opposite side of the bone flap);
4. The subdural effusion cannot be absorbed or has no decreasing trend with conservative treatment and consistent with the indications for surgical treatment;
5. Sign the study informed consent;

Exclusion Criteria:

1. History of craniocerebral disease or craniocerebral surgery;
2. Patients with intracranial infection (cerebrospinal fluid test results must be confirmed by lumbar puncture before inclusion);
3. Combined with ventricular hydrocephalus;
4. Other factors lead to poor prognosis or affect the treatment plan of the patient, even if the effusion can be recovered well, but severe pre-existing disability or severe co-morbidity such as serious heart disease leads to poor prognosis or even death;
5. Pregnant female.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of subdural effusion 1 month after drainage catheter removal. | 1 month after drainage catheter removal.
  The evaluation criteria of whether the effusion has recurred is based on the diagnostic results of the imaging examination. The specific manifestations are that the skull CT examination finds that the effusion has reappeared in the original effusion area.

SECONDARY OUTCOMES:
Incidence of related complications. | 1 month after drainage catheter removal.
  Incidence of related complications (such as intracranial infection and hemorrhage) within 1 month after drainage tube removal.
Method of re-intervention after recurrence of effusion. | 1 month after drainage catheter removal.
  Method of re-intervention after recurrence of effusion (conservative treatment or invasive treatment, specific method).
Length of stay in hospital and detailed economic evaluation. | 1 month after drainage catheter removal.
  Length of stay in hospital and detailed economic evaluation.
GOSE (extended Glasgow Outcome Scale) scores. | 1, 3 and 6 months after drainage catheter removal.
  The primary outcome is indicated by the long-term functional outcomes, including overall mortality and the score on the "Extended Glasgow Outcome Scale" (GOS-E). "Extended Glasgow Outcome Scale" is the unabbreviated scale title, minimum value is 1 and maximum value is 8, which was scored as follows and higher scores mean a better outcome:
  1. death;
  2. persistent vegetative state;
  3. lower severe disability;
  4. upper severe disability (stratum 3 and 4 were considered as severe disability, with permanent requirement for help with daily living);
  5. lower moderate disability;
  6. upper moderate disability (stratum 5 and 6 were considered as mild disability, without a need for assistance in everyday life, that might, however, require special equipment for employment);
  7. lower good recovery;
  8. upper good recovery (stratum 7 and 8 were considered as good recovery).

CONTACTS AND LOCATIONS:
Overall Officials: Jiyao Jiang, Dr., Study Chair — Renji Hospital,School of Medicine,Shanghai Jiao Tong University; Junfeng Feng, Dr., Study Director — Renji Hospital,School of Medicine,Shanghai Jiao Tong University; Qinghua Wang, Dr., Study Director — Southern Medical University, China
Locations (1):
- Brain Injury Center, Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China